CLINICAL TRIAL: NCT01738659
Title: Moderate Versus Low Sodium Diet Intake Effects on Estimated Echocardiographic Pulmonary Capillary Wedge Pressure During 12 Months of Follow up in Compensated Heart Failure Patients.
Brief Title: Estimated Echocardiographic Pulmonary Capillary Wedge Pressure in Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Palermo (Other)
Collaborators: Ospedale G. F. Ingrassia (Other)
Responsible Party: Principal Investigator, Gaspare Parrinello, Associate Professor of Internal Medicine, University of Palermo
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: UNIPA
Record Dates: First submitted 2012-10-23; First posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Heart Failure
Keywords: sodium ,diuretics, PCWP
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- normal sodium diet (120 mmol/die) (Experimental): active comparator: low sodium diet (80 mmol/die)
  Interventions: Dietary Supplement: normal sodium diet

INTERVENTIONS:
Dietary Supplement: normal sodium diet — normal sodium diet (120 mmol/daily) for 1 year

SUMMARY:
The aim of the study was to verify the effects of moderate versus low sodium intake on pulmonary capillary wedge pressure (PCWP), determined by Doppler echocardiography and tissue Doppler imaging in patients suffering from compensated heart failure.

DETAILED DESCRIPTION:
the study outcome is hospital readmission and mortality after 12 months of two different sodium diet.

ELIGIBILITY:
Inclusion Criteria:

* compensated HF patients

Exclusion Criteria:

* decompensated HF patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2008-10; Primary Completion 2010-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
number of hospital readmitted patients | 1 year
  every six months we measure the PCWP by echocardiography

SECONDARY OUTCOMES:
number of death | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: pietro di pasquale, MD, Principal Investigator — G.F. Ingrassia Hospital